CLINICAL TRIAL: NCT01148069
Title: Surgery Combined With IMRT-IGRT in Locally-advanced Prostate Cancers
Brief Title: Surgery Combined With Intensity Modulated Radiation Therapy - Image-Guided Radiation Therapy (IMRT-IGRT) in Locally-advanced Prostate Cancers
Acronym: TARGET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID RCB 2009-A01336-51; LOC/09-07 (Other: Rennes University Hospital); CIC0203/128 (Other: Rennes Clinical Research Center)
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: IMRT-IGRT; radiotherapy toxicity; seminal vesicles
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery combined with IMRT-IGRT (Experimental)
  Interventions: Procedure: Surgery combined with IMRT-IGRT

INTERVENTIONS:
Procedure: Surgery combined with IMRT-IGRT — Patients will have surgery consisting in extensive pelvic dissection and ablation of seminal vesicles. Surgery will be followed by prolonged hormonotherapy (3 years) associated, after 2 months, with prostatic only irradiation.

SUMMARY:
Standard treatment of locally-advanced prostate cancers consists in the association of radiotherapy of prostate and seminal vesicles (SV) and androgen deprivation (AD) for 3 years. This treatment is usually preceded by pelvic lymphadenectomy to assess the possible extension to lymph nodes of prostatic cancer and to avoid irradiating the pelvis in case of no lymph node involvement. However, radiotherapy leads usually to about 30% of grade ≥2 risk of bladder and/or rectal toxicity. This risk particularly depends on the radiation volume. In the aim of lowering the toxicity, the treatment in this study will associate:

* pelvic lymph node dissection and resection of seminal vesicles, allowing decreasing the radiation target volume to the prostate only (and not to irradiate the SV);
* a high-precision radiotherapy technique combining Intensity Modulated Radiation Therapy (IMRT) and Image-Guided Radiation Therapy (IGRT).

DETAILED DESCRIPTION:
This study targets non metastatic prostatic locally-advanced adenocarcinomas which are at high risk of both local progression and metastases. The standard treatment of these tumours associates external beam radiation therapy (EBRT) and 3 years of androgen deprivation (AD) with LH-RH analogue. In the absence of AD and mainly when prostate specific antigen (PSA) is >10 ng/ml, several randomized studies have shown that high doses of EBRT increase biochemical control. Nevertheless, escalating the doses of radiation significantly increases the risk of rectal and/or urinary toxicities. In order to lower the toxicity of irradiation in locally-advanced prostate cancers, and to improve the quality of life of patients, this study aims at decreasing the volume of irradiated healthy tissues. To carry out this objective, we will use a double strategy:

* Limiting the target volume to prostate only by removing seminal vesicles at the time of lymph node dissection,
* Using a technique of high-precision radiation combining Intensity Modulated Radiation Therapy (IMRT) and Image-Guided Radiation Therapy (IGRT).

Based on the literature, we may assume a toxicity rate of 30% during the three years of hormonotherapy with standard treatment (i.e. without removing seminal vesicles). We make the hypothesis of a 20% absolute reduction of toxicity with our protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18,
* Prostate adenocarcinoma (histologically proven),
* Locally-advanced (T3a or Gleason > 7 or PSA ≥ 20 ng/mL),
* Distal half of seminal vesicles unaffected on MRI,
* Non metastatic cancer: negative extension assessment (on prostatic and pelvic MRI and bone scintigraphy),
* Radiotherapy and hormonotherapy indication,
* Medical insurance affiliation,
* Written informed consent.

Non-inclusion criteria:

* Co-morbidity or medical history contraindicating surgery (pelvic lymphadenectomy and seminal vesicle ablation),
* Contraindication to pelvic irradiation,
* Hip prosthesis,
* History of cancer for the last 5 years (except baso-cellular epithelioma),
* History of pelvic irradiation,
* Person deprived of freedom or under guardianship,
* Participation in another biomedical research.

Exclusion Criteria:

* Surgery showing lymph nodes involvement (pelvic radiation indication)
* Surgery without ablation of seminal vesicles
* Surgery with positive margins in seminal vesicles

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-07-30 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Rate of bladder and/or rectal grade ≥2 toxicity (late toxicity) | between 6 months and 3 years
  Rate of bladder and/or rectal grade ≥2 toxicity (CTCAE V4.0) observed between 6 months and 3 years after the beginning of the radiotherapy.

SECONDARY OUTCOMES:
Dose received by the rectum and the bladder with and without seminal vesicles irradiation | Before treatment
  Assessed using a dose-volume histogram
Quality of life | 3 years
  Assessed with EORTC questionnaires (QLQ-C30, QLQ-PR25)
Erectile troubles | 3 years
  Assessed with erectile troubles questionnaire (IIEF-5)
Onset of biological signs evocating a recidive | 3 years
  Assessed with PSA levels
Onset of clinical signs evocating a recidive | 3 years
Specific and global survival | 3 years
Rate of bladder and/or rectal grade ≥2 toxicity (CTCAE V4.0) (early toxicity) | 6 months
  Rate of late bladder and/or rectal grade ≥2 toxicity (CTCAE V4.0) observed 6 months after the beginning of the radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Renaud DE CREVOISIER, MD, PhD, Principal Investigator — Rennes CRLCC Eugène Marquis; Sebastien VINCENDEAU, MD, Study Director — Rennes University Hospital; Eric BELLISSANT, MD, PhD, Study Chair — Rennes University Hospital
Locations (2):
- France (2):
  - Service d'Urologie - Hôpital de Pontchaillou, Rennes
  - Centre Eugène Marquis - CRLCC, Rennes